CLINICAL TRIAL: NCT00529152
Title: A 24-Week, Open Label, Uncontrolled Study of the Safety and Efficacy of Ferriprox™ (Deferiprone) Oral Solution in Iron Overloaded Pediatric Patients With Transfusion-Dependent Anemia
Brief Title: Safety and Efficacy of Ferriprox™ (Deferiprone) Oral Solution in Iron Overloaded Pediatric Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ApoPharma (Industry)
Responsible Party: Dian Shaw, ApoPharma Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LA30-0307
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Results first posted 2009-08-12 (Estimated); Last update posted 2009-09-02 (Estimated); Status verified 2009-08

CONDITIONS: Iron Overload
Keywords: Iron Overload
MeSH Terms: conditions — Iron Overload | interventions — Deferiprone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Other): Ferriprox Oral Solution single treatment
  Interventions: Drug: Deferiprone

INTERVENTIONS:
Drug: Deferiprone — Ferriprox (deferiprone) oral solution will be given orally at a total daily dose of 75 mg/kg body weight or 100 mg/kg body weight, divided into 3 doses, for 24 weeks.
  Other Names: Ferriprox Oral Solution

SUMMARY:
* The primary objective is to assess the safety of Ferriprox oral solution for the treatment of iron overload in pediatric patients with transfusion-dependent anemia.
* The secondary objective is to assess the efficacy of Ferriprox oral solution in reducing iron overload in pediatric patients with transfusion-dependent anemia.

DETAILED DESCRIPTION:
This will be a multi-centre, open label, single treatment, uncontrolled study. A total of 100 iron-overloaded pediatric patients with transfusion-dependent anemia will be enrolled in the study.Eligible patients will receive Ferriprox (deferiprone) oral solution, 100 mg/mL, at a total daily dose of 75 mg/kg body weight or 100 mg/kg body weight, divided in three (3) doses, for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are ≤ 10 years of age.
* Patients who have a confirmed diagnosis of transfusion-dependent anemia, other than Blackfan-Diamond anemia, and have chronic iron overload requiring chelation therapy.
* Patients who are in a chronic transfusion program, and who have received at least eight (8) red blood cell transfusions per year for a minimum of one year.
* Patients who are iron overloaded as assessed by serum ferritin concentration greater than 1000 µg/L.

Exclusion Criteria:

* Patients who have a diagnosis of Blackfan-Diamond anemia.
* Patients who have experienced neutropenia/agranulocytosis (absolute neutrophil count (ANC) < 1.5 x 109/L) or thrombocytopenia (platelet count < 50.0 x 109/L).
* Patients who have had previous treatment with Ferriprox and presented serious adverse reaction or intolerance requiring withdrawal of Ferriprox.
* Patients with evidence of abnormal liver function (ALT level > 3 times the upper limit of normal; entry may be delayed until values return to normal).
* Patients with evidence of renal failure, characterized by serum creatinine level > 2 times the upper limit of normal; entry may be delayed until values return to normal.

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2007-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Mohsen S El Alfy, MD, Principal Investigator — Children Hospital, Ain Shams University, Cairo, Egypt
Locations (4):
- Egypt (2):
  - Abo El Reish Hospital, Cairo University, Cairo
  - Children Hospital, Ain Shams University, Cairo
- Cipto Mangunkusumo National Hospital, Jakarta, Indonesia
- University of Malaya Medical Center, Kuala Lumpur, Malaysia

REFERENCES:
- [Derived] ElAlfy MS, Sari TT, Lee CL, Tricta F, El-Beshlawy A. The safety, tolerability, and efficacy of a liquid formulation of deferiprone in young children with transfusional iron overload. J Pediatr Hematol Oncol. 2010 Nov;32(8):601-5. doi: 10.1097/MPH.0b013e3181ec0f13. PMID 20921906

RESULTS

PARTICIPANT FLOW:
Groups:
- Ferriprox Oral Solution: All subjects were administered Ferriprox Oral Solution three times daily for a total daily dose of either 50, 75 or 100 mg/kg/day. Subjects were initiated at a dose of 50 mg/kg/day, but this dose could be increased after two weeks of therapy depending on the subjects' individual needs.
Period: Overall Study
Arm/Group | Ferriprox Oral Solution
Started | 100
Completed | 95
Not Completed | 5
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ferriprox Oral Solution
Number analyzed (Participants) | 100
Age Continuous [Mean (Standard Deviation); unit: years] | 5.1 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 54
Region of Enrollment [Number; unit: participants]
  Egypt | 76
  Malaysia | 11
  Indonesia | 13
serum ferritin [Mean (Standard Deviation); unit: ug/L] — serum ferritin measures the amount of iron in the blood
  ug/L | 2531.7 (1463.0)

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Adverse Events
Description: Number of Adverse Events over 24 weeks
Time Frame: 24 Weeks
Population: All subjects enrolled (100), had at least one dose of Ferriprox oral solution, all were included in safety analysis
Measure: Number; unit: Adverse Events
Arm/Group | Ferriprox Oral Solution
Number analyzed (Participants) | 100
Adverse Events | 212

2. Secondary Outcome: Change in Serum Ferritin Concentration From Baseline.
Description: The change in serum ferritin concentration from baseline to week 24 was measured and analyzed for all participants in the study
Time Frame: Baseline and 24 weeks
Population: 99 subjects had at least one post baseline measurement of serum ferritin concentration and were eligible for the efficacy analyses in the Intent to Treat population (all subjects). The Last Measurement Carried Forward methodology was used to populate any missing serum ferritin value.
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Ferriprox Oral Solution
Number analyzed (Participants) | 99
ug/L | -355.5 (978.1)
Statistical Analysis 1: Comparison: Ferriprox Oral Solution; Change in Serum Ferritin from baseline to week 24 was compared using regression analysis; null hypothesis was defined as no change in serum ferritin from baseline to week 24; Test type: Superiority or Other; p = 0.0005, Regression, Linear

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right to review manuscript at least 60 days prior to submission and posters/abstracts at least 30 days. If review indicates potentially patentable or confidential information would be disclosed, submission may be delayed an extra 30 days to allow filing the necessary patent applications and to co-operate with the sponsor to protect confidential information. Investigator will delay single center publications until after disclosure of pooled data (all sites) by Sponsor.